CLINICAL TRIAL: NCT00868881
Title: Treatment of Hypertension in Primary Care in Spain
Acronym: TAPAS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Juan Carlos Palma, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-CES-DUM-2008/2
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Hypertension
Keywords: Hypertension; Therapeutic diagnostic attitude; Blood pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: Blood Pressure poorly controlled in the previous year and poorly controlled at the inclusion in the study
- 2: Blood Pressure poorly controlled in the previous year and well controlled at the inclusion in the study.
- 3: Blood Pressure well controlled in the previous year and well controlled at the inclusion in the study
- 4: Blood Pressure well controlled in the previous year and poorly controlled at the inclusion in the study
- 5: Blood Pressure well controlled in the previous year independently of the level of control at the inclusion.
- 6: Blood Pressure poorly controlled in the previous year independently of the level of control at the inclusion.

SUMMARY:
Non-interventional,observational and retrospective study assessing the therapeutic and diagnostic attitude followed in primary care for a hypertensive patient depending on his degree of blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary hypertension and/or treated for hypertension for one year or more
* Clinical data of blood pressure measures for the last 12+/- 2 months before inclusion.

Exclusion Criteria:

* Secondary Hypertension
* Physical or psychological impairment for the understanding of the information to be given to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who has been diagnosed of primary hypertension and/or treated for hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 2160 (Estimated)
Dates: Start 2009-03; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Therapeutic and diagnostic attitude followed in primary care for a hypertensive patient depending on his degree of blood pressure control. | 1 Year

SECONDARY OUTCOMES:
Variation in the Percentage of patients with blood pressure controlled and not controlled during a year of follow-up. | 1 Year
Clinical profile and cardiovascular risk. | 1 Year

CONTACTS AND LOCATIONS:
Locations (167):
- Spain (167):
  - Research Site, A Coruña
  - Research Site, Adeje
  - Research Site, Alacant / Alicante
  - Research Site, Alburquerque
  - Research Site, Alcalá de Henares
  - Research Site, Alcantarilla
  - Research Site, Alfajarín
  - Research Site, Algeciras
  - Research Site, Algimia de Alfara
  - Research Site, Almacelles
  - Research Site, Almería
  - Research Site, Andratx
  - Research Site, ARES (pontedeume)
  - Research Site, Arroyo de la Miel
  - Research Site, As Pontes de García Rodríguez
  - Research Site, Avilés
  - Research Site, Águilas
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Barreiros (casco Urbano)
  - Research Site, Belmonte
  - Research Site, Beniarjó
  - Research Site, Bilbao
  - Research Site, Boiro (boiro)
  - Research Site, Boqueixon (ponteulla)
  - Research Site, Burgos
  - Research Site, Burjassot
  - Research Site, Cadiz
  - Research Site, Calahorra
  - Research Site, Calamonte
  - Research Site, Calatayud
  - Research Site, Caldes de Montbui
  - Research Site, Campanario
  - Research Site, Carballo (carballo)
  - Research Site, Castalla
  - Research Site, Castellon
  - Research Site, Ceuta
  - Research Site, Cieza
  - Research Site, Corbera de Llobregat
  - Research Site, Corme-Porto
  - Research Site, Córdoba
  - Research Site, Cubells
  - Research Site, Cuenca
  - Research Site, Cullera
  - Research Site, Dacón
  - Research Site, Don Benito
  - Research Site, Dos Hermanas
  - Research Site, El Bonillo
  - Research Site, El Ejido
  - Research Site, el Pla del Penedès
  - Research Site, ELX / Elche
  - Research Site, Fraga
  - Research Site, Fraile
  - Research Site, Fuente del Arco
  - Research Site, Gallarta
  - Research Site, Gallur
  - Research Site, Gandia
  - Research Site, Gavà
  - Research Site, Gáldar
  - Research Site, Getafe
  - Research Site, Getxo
  - Research Site, Gijón
  - Research Site, Girona
  - Research Site, Godella
  - Research Site, Grado
  - Research Site, Granada
  - Research Site, Granollers
  - Research Site, Guía de Isora
  - Research Site, Higuera la Real
  - Research Site, Jerez de la Frontera
  - Research Site, La Línea de la Concepción
  - Research Site, La Orotava
  - Research Site, La Pesga
  - Research Site, Las Palmas de Gran Canaria
  - Research Site, Las Torres de Cotillas
  - Research Site, Leganés
  - Research Site, Legutio
  - Research Site, León
  - Research Site, Lestrobe
  - Research Site, Linyola
  - Research Site, Lora del Río
  - Research Site, Los Corrales de Buelna
  - Research Site, Los Realejos
  - Research Site, Los Yébenes
  - Research Site, Madrid
  - Research Site, Madroñera
  - Research Site, Manises
  - Research Site, Manresa
  - Research Site, Marmolejo
  - Research Site, Málaga
  - Research Site, Miranda de Ebro
  - Research Site, Mislata
  - Research Site, Mollet del Vallès
  - Research Site, Monforte del Cid
  - Research Site, Monistrol de Montserrat
  - Research Site, Monover/monovar
  - Research Site, Montilla
  - Research Site, Morata de Jalón
  - Research Site, Mutxamel
  - Research Site, Nava de la Asunción
  - Research Site, Navalperal de Pinares
  - Research Site, Noreña
  - Research Site, Olivenza
  - Research Site, Onil
  - Research Site, Palau-saverdera
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Parets del Vallès
  - Research Site, Petrel
  - Research Site, Pinto
  - Research Site, Pizarra
  - Research Site, Porreres
  - Research Site, Portals Nous
  - Research Site, Posada de Llanes
  - Research Site, Pozo-Cañada
  - Research Site, Puerto Lumbreras
  - Research Site, Purias
  - Research Site, Quart de Poblet
  - Research Site, Quintana de la Serena
  - Research Site, Quiroga (casco Urbano)
  - Research Site, Roturas
  - Research Site, Sabadell
  - Research Site, San Martín de Luiña
  - Research Site, San Vicente de Alcántara
  - Research Site, Sant Carles de la Ràpita
  - Research Site, Sant Cugat Sesgarrigues
  - Research Site, Sant Feliu de Llobregat
  - Research Site, Sant Martí Sarroca
  - Research Site, Santa Coloma de Gramenet
  - Research Site, Santander
  - Research Site, Segorbe
  - Research Site, Serradilla
  - Research Site, Seville
  - Research Site, Son Ferriol
  - Research Site, Soto de la Marina
  - Research Site, Taboadela
  - Research Site, Tauste
  - Research Site, Toledo
  - Research Site, Tordesillas
  - Research Site, Torre de Don Miguel
  - Research Site, Torredelcampo
  - Research Site, Torrejoncillo
  - Research Site, Torrejón de Ardoz
  - Research Site, Torrellano
  - Research Site, Torres de Segre
  - Research Site, Torrevieja
  - Research Site, Trapagaran
  - Research Site, Tui
  - Research Site, Utrillas
  - Research Site, Valencia
  - Research Site, Valencia de Alcántara
  - Research Site, Valladolid
  - Research Site, Vallirana
  - Research Site, Vigo
  - Research Site, Viladecans
  - Research Site, Vilanova (lourenza)
  - Research Site, Villafranca de los Barros
  - Research Site, Villagonzalo-Pedernales
  - Research Site, Villalba de los Barros
  - Research Site, Vitoria-Gasteiz
  - Research Site, Xàtiva
  - Research Site, Xinzo de Limia
  - Research Site, Yecla
  - Research Site, Zafra
  - Research Site, Zalamea de la Serena
  - Research Site, Zamora
  - Research Site, Zaragoza